CLINICAL TRIAL: NCT00479440
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SAM-315 Administered Orally to Healthy Adult Subjects
Brief Title: Study Evaluating the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of SAM-315 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3182A1-100
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-(naphthalen-1-ylsulfonyl)-5-(piperazin-1-yl)-1H-indazole

INTERVENTIONS:
Drug: SAM-315

SUMMARY:
To assess the safety and tolerability of ascending single oral doses of SAM-315, an investigational drug, in healthy adult subjects. To obtain a preliminary pharmacokinetic (PK) and pharmacodynamic (PD) profiles of SAM-315 in healthy subjects and to evaluate the effect of a high-fat meal on the PK of SAM-315, an investigation drug, administered to healthy adult subjects.

ELIGIBILITY:
Inclusion criteria:

* Men and women of nonchildbearing potential aged 18 to 45 years
* Body mass index in the range of 18 to 30 kg/m2 and body weight ≥50 kg.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and digital 12-lead electrocardiogram (ECG). Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and creatinine levels must be within the upper limit of normal for eligibility.

Exclusion criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Any clinically important deviation from normal limits in physical examination, vital signs, digital 12-lead ECGs, or clinical laboratory test results.
* Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) or alcoholic beverages within 48 hours and, grapefruit, grapefruit-containing products is prohibited 72 hours before study day 1.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56
Dates: Start 2006-08; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer